CLINICAL TRIAL: NCT03493633
Title: Study of Use of the EzyGain Training and Rehabilitation Device for Walking at Home
Brief Title: Use EzyGain at Home (Device for Walking at Home)
Acronym: EzyGain
Status: Terminated | Type: Observational
Why Stopped: early termination - fault of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P170705J; 2017-A03170-53 (Other: IDRCB)
Record Dates: First submitted 2018-03-01; First posted 2018-04-10 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Physical Disability; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EzyGain at Home: Setting up a walking device at home for people aged 60 years with partial walking disability regardless of etiology and pathology leading to walking disability.
  Interventions: Device: EzyGain

INTERVENTIONS:
Device: EzyGain — Each patient performs a minimum of 3 sessions per week with the investigator / APA investigator, for 4 weeks, each walk for a few minutes (<60 min).
  Evaluation of the spontaneous physical activity of the patient by actimetry for seven days QAPPA (questionnaire of physical activity for elderly person) a week and a month after the training phase of four weeks

SUMMARY:
Our research hypothesis is that the practice of walking on a secure treadmill is possible at home and allows the patient to increase the training work of walking in everyday life compared to a conventional care.

DETAILED DESCRIPTION:
Our research hypothesis is that the practice of walking on a secure treadmill is possible at home and allows the patient to increase the work of training of walking in everyday life compared to a conventional care. In addition, we believe that this practice should be supervised by a caregiver trained by the physiotherapist / APA investigator, in order to increase the use of the device.

The people concerned by this protocol are those who have a partial disability of walking whatever the pathology and the underlying deficiencies.

Main objective: To evaluate the feasibility of using EzyGain at home.

Main Evaluation Criteria: Number of sessions performed on the device during the duration of the study, compared to the number of scheduled sessions.

Secondary objectives

Secondary objective 1: make a partial transfer of the supervision of the physiotherapist / APA investigator's sessions to the caregiver.

Secondary Objective 2: To evaluate whether the exercise period on the device increases the amount of spontaneous physical activity of the patient after the end of the period compared to the average spontaneous physical activity prior to the exercise period.

Population concerned:

Population over 60 years of age with partial walking disability regardless of etiology and pathology leading to walking disability.

Population coming into consultation in the services of Dr. Teixeira and Pr. Yelnik of GH Saint Louis Lariboisière Fernand Widal.

Partial incapacity of walking. Availability at home during their participation period (weeks of walking exercise + weeks of evaluation of physical activity).

Ethnicity indifferent Indifferent sex Patient with a close volunteer caregiver to participate in the study and receive training from the investigator / APA investigator and then manage sessions autonomously.

Anyone who would like to train more regularly on the walk and at home because unable to go out.

Who uses or does not use technical assistance to walk or move Patient who falls or is at risk of falling and, as a result, limits his progress.

Possibility of installation of the device in the patient's home. Patient affiliated to a social security scheme

Practical sequence:

Selection and medical inclusion of the patient by one of the investigating physicians and delivery of consent. During this visit, the doctor judges the eligibility criteria, explains the research to the patient, gives him the informed consent that is signed on the spot.

Among the eligibility criteria, there must be a caregiver close to the patient, who is willing to participate in the research. If he is present during this visit, he signs his consent to participate in the research. If he is absent during this visit, the patient gives his coordinates, the doctor calls him to explain the research, and sends his consent by mail, which the caregiver returns signed by mail to the doctor. It only remains to verify that the apartment can accommodate the device EzyGain.

Evaluation of the accessibility of the home by the EzyGain team. If the apartment can accommodate the device, then the patient is included in the search. If the apartment can not accommodate the device, then the patient is not included.

The first visit takes place on site with the investigator / APA investigator and an investigator. Laying the Actigraph ©.

Evaluation of the spontaneous physical activity of the patient by actimetry for seven days + QAPPA (questionnaire of physical activity for old person).

Beginning of the training phase on the device. The dosage of the activity (frequency of sessions and practical content) and the possibility of supervising additional sessions by a family caregiver is determined by the investigating physiotherapist / APA investigator.

Each patient performs a minimum of 3 sessions per week with the investigator / APA investigator, for 4 weeks, each walk for a few minutes (<60 min).

Evaluation of the spontaneous physical activity of the patient by actimetry for seven days QAPPA (questionnaire of physical activity for elderly person) a week and a month after the training phase of four weeks

ELIGIBILITY:
Inclusion Criteria:

* Person over the age of 60
* Availability at home during their participation period (walking exercise weeks + physical activity assessment weeks).
* Patient with a volunteer close caregiver to participate in the study and receive training from the investigator/APA investigator and then manage autonomy sessions.
* Person who would like to train more regularly in the walk and at home because unable to get out. Person who uses or does not use technical assistance to walk or move
* Person in a State to sign informed consent alone
* Possibility of installation of the device in the patient's home (the dimensions of the lift/doors/parts allow the device to be entered in the apartment, as well as not to hinder the daily life of the patient too heavily).
* Patient affiliated with a Social security plan
* Person who has a partial limitation of walking activity (partial inability to walk) and in whom, re-education of walking is relevant to improve performance (whether or not the patient does this re-education at the time of the visit of selection). The criteria for limiting walking activity are:
* Speed limitation
* Endurance limitation
* Limitation of the operating perimeter
* Limitation of the dynamic balancing during walking failure to position the foot or feet during walking
* Falls
* Availability at home during their time of participation.
* Indifferent ethnic origin
* Indifferent sex

Exclusion Criteria:

* Uncontrolled heart failure
* Uncontrolled respiratory insufficiency
* Uncontrolled coronary insufficiency
* Impossibility of installing the device at home
* Severe cognitive impairment with risk of using the device alone, outside of the instructions
* Absence of a caregiver to follow a continuous training of the physiotherapist / - APA investigator to supervise independently one or two sessions per week

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population over 60 years of age with partial walking disability regardless of etiology and pathology leading to walking disability.
  Population coming into consultation in the services of Dr. Teixeira and Pr. Yelnik of GH Saint Louis Lariboisière Fernand Widal.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Number of sessions performed on the device during the duration of the study | Up to 4 weeks
  Count of the number of sessions performed. A session is considered to be performed when the patient is walking for at least one minute on the EzyGain treadmill with the APA investigator / caregiver.

SECONDARY OUTCOMES:
Number of sessions performed autonomously by the caregiver | Up to 4 weeks
  Measure of the number of self-help sessions performed by the caregiver and their proportion to the total number of sessions completed.
Physical activity evaluate by actimetry before the training period | At days 7 before the training period
  Evaluate spontaneous physical activity by actimetry over a continuous period of 7 days before the beginning of the exercise period.
  At day #1 of the 7-day period : put the Actigraph© on the patient At day #7 of the 7-day period : take the Actigraph© off the patient
Physical activity evaluate by QAPPA before the training period | At days 7 before the training period
  Evaluate spontaneous physical activity by QAPPA, 7 days before the beginning of the exercise period.
  At day #7 of the 7-day period do the QAPPA
Physical activity evaluate by actimetry just after the training period | At days 7 after the end of the training period
  Evaluate spontaneous physical activity by actimetry over a continuous period of 7 days starting the day after the end of the exercise period.
  At day #1 of the 7-day period : put the Actigraph© on the patient At day #7 of the 7-day period : take the Actigraph© off the patient
Physical activity evaluate by QAPPA just after the training period | At days 7 after the end of the training period
  Evaluate spontaneous physical activity by QAPPA over period of 7 days starting the day after the end of the exercise period.
  At day #7 of the 7-day period do the QAPPA
Physical activity evaluate by actimetry 3 weeks after the training period | At 3 weeks after the training period
  Evaluate spontaneous physical activity by actimetry over a continuous period of 7 days starting 3 weeks after the end of the exercise period.
  At day #1 of the 7-day period : put the Actigraph© on the patient At day #7 of the 7-day period : take the Actigraph© off the patient
Physical activity evaluate by QAPPA 3 weeks after the training period | At 3 weeks after the training period
  Evaluate spontaneous physical activity by QAPPA over a continuous period of 7 days starting 3 weeks after the end of the exercise period.
  At day #7 of the 7-day period do QAPPA

CONTACTS AND LOCATIONS:
Overall Officials: Alain YELNIK, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Physique et de Réadaptation - Hôpital F.Widal, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided